CLINICAL TRIAL: NCT00969293
Title: An Open-label, Dose Escalating Study to Assess the Safety and Tolerability of a Single Administration of FOV2302 (Ecallantide) in Patients With Macular Edema Associated With Central Retinal Vein Occlusion
Brief Title: Study to Assess the Safety and Tolerability of a Single Administration of FOV2302 (Ecallantide) in Patients With Macular Edema Associated With Central Retinal Vein Occlusion
Acronym: FOV2302
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Fovea Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOV2302/CLIN/101/P
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Macular Edema; Central Retinal Vein Occlusion
Keywords: Macular Edema; Occlusive retinal vascular disease; Central Retinal Vein Occlusion; CRVO
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — ecallantide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: FOV2302 (Ecallantide) — Single intravitreal injection into the relevant eye.
  Five dose levels will be studied from 5 to 90µg and a maximum of 6 subjects will be included at each dose level.
  Duration of Treatment: Single injection with 3 months follow-up.

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of a single administration of FOV2302 (ecallantide) in patients with macular edema associated with central retinal vein occlusion.

DETAILED DESCRIPTION:
Occlusive retinal vascular disease is not uncommon. Central retinal vein occlusion (CRVO) is the second most common vision-impairing vascular disorder of the retina following diabetic retinopathy. Severe visual loss from CRVO is caused by a combination of retinal edema and neovascular proliferation and ischemia. Vascular endothelial factors as they stimulate angiogenesis and increase vascular permeability, are majors pathogenic factors in CRVO. Counteracting these neovascular effects provide significant therapeutic benefit to subjects suffering from this disorder. Macular edema in this condition results from a conjunction of several, as yet, partially unknown factors.

Macular edema may occur in diseases causing cumulative injury over many years, such as diabetic retinopathy, or as a result of more acute events, such as branch retinal vein occlusion (BRVO) or central retinal vein occlusion (CRVO).

ELIGIBILITY:
Inclusion Criteria:

* Recent onset (< 6 months), non-ischemic CRVO (defined as association of documented retinal hemorrhage in all 4 quadrants of the retina with dilated veins) in patients who have not received treatment for their condition (e.g., no periocular depot or intraocular treatment [including corticosteroid and anti-VEGF], systemic corticosteroids or laser nor hemodilution).
* Retinal thickness measured by Stratus OCT > 250µm in the central subfield of study eye at baseline.
* BCVA score (measured by the ETDRS chart between 5 letters (20/800 Snellen equivalent) and 65 letters (20/50) in the study eye at baseline.
* Media clarity, pupillary dilation and participant cooperation sufficient for adequate fundus photographs.
* Females of childbearing potential using adequate birth control at Day 0 until study completion.
* Patient able (in the opinion of the investigator) and willing to return for all scheduled visits and assessments.
* Ability to read, understand and willingness to provide informed consent.

Exclusion Criteria:

* Rubeosis iridis or neovascular glaucoma at baseline.
* Preretinal neovascularisation at baseline.
* Ischemic CRVO, defined by more than 10 disc area of non-perfusion on fluorescein angiography at baseline.
* Any grade of diabetic retinopathy.
* Other eye condition that could contribute to macular edema or cause retinal vascular changes (including vitreomacular traction, uveitis and inflammatory disease, etc).
* Patients who have received treatment for their condition (e.g., no periocular depot or intraocular treatment [including corticosteroid and anti-VEGF], systemic corticosteroids or laser nor hemodilution).
* Ocular surgery (including cataract extraction, scleral buckle, etc.) and/or YAG capsulotomy within 3 months preceding treatment date or anticipated within the 3 months following treatment administration.
* Poorly controlled ocular hypertension and/or glaucoma (IOP greater than 25 mmHg despite maximal therapy).
* History of pars plana vitrectomy.
* Aphakia or anterior chamber intraocular lens.
* Presence of visible sclera thinning or ectasia.
* Presence of substantial cataract or other media opacity that, in the opinion of the investigator, is likely to interfere with visualization of the fundus or completion of study measurements.
* Any active ocular or peri-ocular infection (including conjunctivitis, chalazion or significant blepharitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability parameters to determine MTD: 1. Systemic parameters: adverse events (AEs), coagulation parameters (APTT, ACT) 2. Ophthalmologic parameters: BCVA, OCT, ocular inflammation, IOP | 3 months post-dose

SECONDARY OUTCOMES:
Assess the pharmacodynamics up to five dose levels of a single administration of FOV2302 (ecallantide) by longitudinal measurements of the percent change of the macula thickness versus baseline as measured by OCT | 3 months post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Alain Gaudric, MD, Study Chair — Hopital Lariboisiere
Locations (8):
- France (8):
  - CHU d'Amiens, Centre Saint-Victor, Amiens
  - Centre Intercommunal de Creteil, Créteil
  - CHU de Dijon, Hôpital Général, Dijon
  - Clinique Monticelli, Marseille
  - CHU de Nantes, Nantes
  - Centre Hospitalier National d'Ophthalmologies des XV-XX, Paris
  - Hopital Lariboisiere, Paris
  - Fondation Rothschild, Paris